CLINICAL TRIAL: NCT04792164
Title: Effect of Ultra-Sound Guided Pre-emptive Nerve Block on Post-operative Pain Following Open Inguinal Hernia Repair: Randomised Control Trial
Brief Title: Effect of Ultra-Sound Guided Pre-emptive Nerve Block on Post-operative Pain Following Open Inguinal Hernia Repair.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Nasser Mohamed Amer, Assistant professor of General Surgery in Imam Abdulrahman bin Faisal University, Imam Abdulrahman Bin Faisal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: USG-PENB-IHR
Record Dates: First submitted 2021-02-09; First posted 2021-03-10 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Intervention Model Description: 2 Arms
  Arm1) The experimental group will receive US guided nerve block by Lidocaine+Marcaine concentration (1%+.25%).
  Arm2) The control group will receive usual infiltration by Lidocaine+Marcaine concentration (1%+.25%).
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blinded ( Patient and researcher recruiter)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental group will receive US guided nerve block (Experimental): The experimental group will receive US guided nerve block by lidocaine before open inguinal hernia repair.
  Interventions: Procedure: Ultra sound guided nerve block
- The control group will receive usual infiltration (Other): The control group will receive usual infiltration by lidocaine before open inguinal hernia repair.
  Interventions: Procedure: Usual infiltration

INTERVENTIONS:
Procedure: Ultra sound guided nerve block — Ultra sound guided nerve block by lidocaine before open inguinal hernia repair.
  Arms: The experimental group will receive US guided nerve block
Procedure: Usual infiltration — Usual infiltration by lidocaine before open inguinal hernia repair.
  Arms: The control group will receive usual infiltration

SUMMARY:
A hernia occurs when an organ 'like intestines' or fatty tissue protrude through a weak point in muscle or connective tissue and one of the most common types of hernia is inguinal. Inguinal hernia defined as a bulge in the inguinal region or scrotum, may be accompanied by dull or burning pain, which worsens by exercise or cough. There are 2 types of inguinal hernia: direct and indirect. Direct inguinal hernia occurs because of a defect or weakness in the transversalis fascia area of the Hesselbach triangle. On the other hand, the indirect inguinal hernia which is the most common inguinal hernia follows the tract of inguinal canal and result from a persistent processus vaginalis.

Immediate pain after inguinal herniorrhaphy delays the ambulation which leads to delay in the hospital discharge. Besides that, is the chronic pain that affect 50% of patients which is an important issue that needs to be dealt with.

Our aim of this study, is to compare between postoperative period in the patients who received US guided nerve block and in patients who received infiltration only before open inguinal hernia repair, and to show that pre-emptive local anaesthesia will result in better pain control, less postoperative complication, earlier mobilisation, earlier recovery and less analgesia consumption by patients.

DETAILED DESCRIPTION:
In this study our aim in detail is to:

1. Asses the outcomes (early postoperative pain management in day case "day 1,2,3, 30 and 3 month and 6 month" , length of hospital stay, analgesia consumption، recovery to work, driving and usual activity) of the US guided nerve block in patients who underwent inguinal hernia repair comparing to patient who received only skin infiltration.
2. Evaluate the advantages of the US guided nerve block in postoperative inguinal hernia repair patients.
3. Demonstrate its compatibly as a one day procedure (less length of hospital stay), with earlier return to work and driving and recovery in general.
4. Compare our result with other international studies result.

Study in details:

it is Randomised Control Trial, Double blinded (patients and recruiter), study will be conducted in King Fahd University Hospital, Khobar, Eastern Province, Saudi Arabia. It contains 2 Arms ,Two Parallel groups. The experimental group will receive US guided nerve block and the control group will receive usual infiltration. Lidocaine+ Marcaine will be used in both group with same concentration (1%+.25%). The random allocation will be done using simple random allocation with a help of the following software (random.org).

Will compare the two groups regarding, a questionary with visual analogue will be distributed and data will be collected by recruiters regarding pain scale, length of hospital stay, return to work, return to driving and usual activity, and analgesia consumption post operative, all in day 1,2,3,4,30,3 month and 6 month post operatives (details in outcome section).

We are expecting to have a reduction in pain score from severe to moderate, about 20% in experimental group, and reducing the length of hospital stay from 1-2 days to one day procedure. And reduction in consumption of Analgesia postoperative.

our sample size will be 134 with a power of 80% and an effect size of 0.5, will include all patients who will have inguinal hernia repair and meet our inclusion criteria, in period of 12-18 months starting after obtaining of IRB approval.

* Inclusion criteria:

  1. Patients who underwent elective inguinal hernia repair (will consider the hernia size).
  2. Age from 18-70.
  3. Their ASA score 1,2 or 3 (American Society of Anesthesia)
  4. Operation under general anaesthesia.
  5. Open inguinal hernia repair.
* Exclusion criteria:

  1. All emergency inguinal hernia repair and recurrent hernia.
  2. Children and pregnant women.
  3. Patients having regional anaesthesia. (Spinal/Local).
  4. Laparoscopic inguinal hernia.

Data Management and analysis plan:

* SPSS latest version will be used for data analysis.
* Summary statistic will be obtained as frequency, and percentage for qualitative data, and means, medians and standard deviations from continuous variables.
* Analysis will be done by epidemiologist and biostatistician.

Ethical Considerations:

* Our study does not have any physical, psychological, social, legal, economic risk.
* The study will be reviewed by IRB, ethics committee; then the approval will be obtained.
* Written approval will be obtained from the patients prior to the procedure.
* Preemptive analgesia and infiltration are usually used in our practice and aim to compare.

ELIGIBILITY:
* Inclusion criteria:

  1. Patients who underwent elective inguinal hernia repair (will consider the hernia size).
  2. Age from 18-70. (70 with no other comorbiditeis)
  3. Their ASA score 1,2 or 3 (American Society of Anesthesia)
  4. General Anesthesia.
  5. Open inguinal hernia repair.
* Exclusion criteria:

  1. All emergency inguinal hernia repair and recurrent hernia.
  2. Children and pregnant women.
  3. Patients having regional anesthesia. (Spinal/Local).
  4. Laparoscopic inguinal hernia.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-12-29 (Estimated); Study Completion 2023-06-29 (Estimated)

PRIMARY OUTCOMES:
Pain Scale (from 1 to 10) 1 is the minimum and 10 the maximum pain severity. | Day 1 postoperative.
  Assessment of pain scale post operative, lower score mean a better outcome.
Pain Scale (from 1 to 10) 1 is the minimum and 10 the maximum pain severity. | Day 2 postoperative.
  Assessment of pain scale post operative, lower score mean a better outcome.
Pain Scale (from 1 to 10) 1 is the minimum and 10 the maximum pain severity. | Day 3 postoperative.
  Assessment of pain scale post operative, lower score mean a better outcome.
Pain Scale (from 1 to 10) 1 is the minimum and 10 the maximum pain severity. | Day 4 postoperative.
  Assessment of pain scale post operative, lower score mean a better outcome.
Pain Scale (from 1 to 10) 1 is the minimum and 10 the maximum pain severity. | Day 30 postoperative.
  Assessment of pain scale post operative, lower score mean a better outcome.
Pain Scale (from 1 to 10) 1 is the minimum and 10 the maximum pain severity. | 3 month postoperative for chronic pain.
  Assessment of pain scale post operative, lower score mean a better outcome.
Pain Scale (from 1 to 10) 1 is the minimum and 10 the maximum pain severity. | 6 month postoperative for chronic pain.
  Assessment of pain scale post operative, lower score mean a better outcome.
Assessment of early mobilisation. | Day 1 postoperative period.
  When the patient started to mobilise? assessed by monitoring the patients postoperative and record when he started to mobilise.
Assessment of early mobilisation. | Day 2 postoperative period.
  When the patient started to mobilise? assessed by monitoring the patients postoperative and record when he started to mobilise.
Assessment of early mobilisation. | Day 3 postoperative period.
  When the patient started to mobilise? assessed by monitoring the patients postoperative and record when he started to mobilise.
Retain to driving (how many days between surgery and patient back to dive) | Postoperative period up to 8 weeks.
  When the patient back to drive his car? assessed by monitoring the patients postoperative and record when he started to drive the car again.
Retain to work (how many days between surgery and patient back to his work) | Postoperative period up to 8 weeks.
  When the patient back to his work or usual activity? assessed by monitoring the patients postoperative and record when he started to work again.
Length of hospital stay (in days). | immediately after the surgery until patient discharged.
  Length of hospital stay post open inguinal hernia repair ( how many days patient spend in the hospital postoperative).
Frequency of analgesia consumption postoperative. | Day 1 postoperative.
  Analgesia consumption by patient postoperative (How frequent patient taking analgesia postoperative).
Frequency of analgesia consumption postoperative. | Day 2 postoperative.
  Analgesia consumption by patient postoperative (How frequent patient taking analgesia postoperative).
Frequency of analgesia consumption postoperative. | Day 3 postoperative.
  Analgesia consumption by patient postoperative (How frequent patient taking analgesia postoperative).
Frequency of analgesia consumption postoperative. | Day 4 postoperative.
  Analgesia consumption by patient postoperative (How frequent patient taking analgesia postoperative).
Frequency of analgesia consumption postoperative. | Day 5 postoperative.
  Analgesia consumption by patient postoperative (How frequent patient taking analgesia postoperative).
Frequency of analgesia consumption postoperative. | Day 6 postoperative.
  Analgesia consumption by patient postoperative (How frequent patient taking analgesia postoperative).
Frequency of analgesia consumption postoperative. | Day 7 postoperative.
  Analgesia consumption by patient postoperative (How frequent patient taking analgesia postoperative).